CLINICAL TRIAL: NCT03675594
Title: Retention of Computer Aided Design and Computer Aided Manufacturing Titanium Versus Cobalt/Chromium Maxillary Single Denture Bases: A Randomized Clinical Trial.
Brief Title: Retention of Computer Aided Design and Computer Aided Manufacturing Titanium Versus Co/Cr Single Dentures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Gamal Ismail Mohamed, Assistant lecturer of prosthodontics, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 28912240102212
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Edentulous Mouth
Keywords: Dislodgement force; Digital denture; CAD/CAM metallic dentures
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the participants will not be told which type they received till obtaining the final results of both types.Outcomes will be collected only by the supervisor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention arm (Experimental): the group of participants will take the CAD/CAM titanium denture bases and assessment during and after the first 3 months after delivery of the first type.
  Interventions: Device: CAD/CAM titanium denture base
- intervention arm 2 (Experimental): the same group of participants will take the CAD/CAM cobalt/chromium denture bases and assessment during and after the second 3 months after delivery of the second type.
  Interventions: Device: CAD/CAM cobalt/chromium denture bases

INTERVENTIONS:
Device: CAD/CAM titanium denture base — metallic denture base made of titanium
  Arms: intervention arm
Device: CAD/CAM cobalt/chromium denture bases — metallic denture bases made of cobalt/chromium
  Arms: intervention arm 2

SUMMARY:
* Steps in short: Undergoing the conventional steps of maxillary single denture construction till the step of framework construction that will be designed and constructed using CAD/CAM after optical scanning of the master cast ( 2 frameworks to cover the palate and crest of the ridge : one made of titanium and the other made of cobalt/chromium) then conventional steps will be undergone including bite, Try-in and delivery ending by measuring the denture retention.
* Number of visits & follow up period :

Visits: will be 5-6 visits for each patient. Follow up period: 6.5 months (immediately post-insertion then after 1 week then after 3 months for the first type then 2 weeks washout period and the same for the second type)

DETAILED DESCRIPTION:
The study will be carried out in the department of prosthodontics-cairo university. Patients will be selected from the out-patient clinic according to the inclusion criteria, The primary impression will be made with alginate (cavex-normal set) and will be border-molded to get the acceptable extension and border thickness, a tray will be prepared with self-activated acrylic resin over the study cast. A secondary impression will be made with heavy putty consistency as a border molding material and the final impression will be made with light rubber base (3M) impression material, Then Pouring of the final impressions with type 4 Hydrocal dental stone (Hydrocal Dental stone, Bayer, and Germany). Master casts will be optically scanned using 3 shape optical scanner. Duplication of master casts will be done using silicone duplicating material. Titanium and cobalt/chromium metallic bases will be milled using 3shape milling machine to cover the palate with mesh extension over the ridge. They will be tried intra-orally regarding sitting and stability. Occlusal rim will be set on titanium metallic base then face bow record will be recorded then mounting the maxillary master cast. Centric relation will be registered then mounting of the mandibular cast will be done. The same will be done for the duplicate cast with the Cobalt/Chromium metallic base. Then Setting of the anatomical teeth for both master casts then try-in stage will be checked intra-orally then packing of cast and duplicate cast with conventional heat cured acrylic resin (Dentsply, Dentsply limited, Weybridge, Surrey. England) after flasking each denture will be finished.

The dentures will be delivered, then the assessment will be immediately and after 1 week then after 3 months that a hook screw with its nut (Digital force gauge instrument, model 475044) will be secured in the polished mid-palatal surface of the upper denture using metallic adhesive to record the amount of the force required for dislodgment. The pull end of the digital force gauge device will be connected to the hook positioned at maxillary dentures for one type of the two dentures and will be pulled vertically until denture dislodgement occurred, then the patient will take off his first type of denture for 2 weeks as a washout period then the second type of denture will be delivered and the same assessment will be done.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous maxillary arch and fully dentate mandibular arch with adequate interarch space.
* The edentulous ridges should be covered by firm healthy mucosa.
* Angle class I maxillomandibular relationship
* Healthy and co-operative patients.

Exclusion Criteria:

* Patients with bad habits as severe clenching or bruxism, drug or alcohol addiction, moderate or heavy smoking (greater than I 0 cigarettes/day).
* Previous history of radiotherapy or chemotherapy.
* Any skeletal problem dictates surgical intervention.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Retention of single denture | 6.5 months
  the dislodgement force of the denture will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: iman rady, professor, Study Director — head of evidence based dentistry
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Manyal, Egypt

IPD SHARING:
Plan to Share IPD: No
it will not be shared with other researchers except my supervisor